CLINICAL TRIAL: NCT03956095
Title: Preoperative Nutrition Intervention for Patients Undergoing Primary Surgical Debulking of Ovarian Cancer: A Feasibility Study
Brief Title: Study of Nutritional Supplement Shakes in People About to Receive Their Debulking Surgery for Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-108
Record Dates: First submitted 2019-05-17; First posted 2019-05-20 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Debulking Surgery for Ovarian Cancer
Keywords: Nutritional Supplement Shakes; 19-108

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ensure Surgery Immunonutrition Shake supplements: Participants will be provided with and instructed to drink three Ensure Surgery Immunonutrition Shake supplements per day for seven days prior to their scheduled procedure.
  Interventions: Dietary Supplement: Ensure Surgery Immunonutrition Shake supplements; Other: Daily Food Intake form

INTERVENTIONS:
Dietary Supplement: Ensure Surgery Immunonutrition Shake supplements — Three Ensure Surgery Immunonutrition Shake supplements per day for seven days prior to their scheduled procedure.
Other: Daily Food Intake form — On the day of surgery, the patient will return her Daily Supplement/Food Intake Forms and complete the Day of Surgery Intake Form can also be completed the day before surgery and the Daily Supplement/Food Intake Forms can be returned at the patient's postoperative appointment.

SUMMARY:
The purpose of this study is to find out if it is possible to establish a nutritional support program for people who are scheduled to receive primary debulking surgery.

Design: This will be a prospective observational study to assess the feasibility of implementing a preoperative nutrition supplementation program.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Scheduled to undergo primary surgical debulking of ovarian, fallopian tube and primary peritoneal cancer
* Have a sufficient preoperative window during which the intervention can occur, with the last day of supplementation at least one and no more than two days prior to surgery; scheduling of the procedure should not be delayed due to participation in this investigation

Exclusion Criteria:

* Have received neoadjuvant chemotherapy
* Debulking surgery scheduled less than 8 days from initial visit
* Are scheduled for a minimally invasive procedure
* Unable to tolerate oral intake or have gastrointestinal issues that would prevent or prohibit oral supplement consumption
* Have diabetes mellitus
* Have allergies to the Ensure Surgery Immunonutrition Shake supplement
* Have galactosemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian Cancer
Study Population: Eligible patients will include those who present to MSK for primary surgical management of ovarian cancer.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
rate of patient participation | 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vance Broach, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Baptist Alliance MCI, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm